CLINICAL TRIAL: NCT00291616
Title: A Multicenter, Randomized, Controlled Trial of Combination Therapy for HBeAg Positive Chronic Hepatitis B: Comparing Thymosin Alpha 1 and Pegylated Interferon-alpha2a With Pegylated Interferon-alpha2a Alone.
Brief Title: Efficacy Study of Thymosin alpha1 & Pegylated Interferon-alpha2a to Treat Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Roche Pharma AG (Industry); SciClone Pharmaceuticals (Industry)
Responsible Party: Won Kim, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-05-008
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Hepatitis B
Keywords: chronic hepatitis B, pegylated interferon, thymosin alpha
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Pegylated Interferon-alpha2a
  Interventions: Drug: Pegylated Interferon-alpha2a
- 2 (Active Comparator): Thymosin alpha1 & Pegylated Interferon-alpha2a
  Interventions: Drug: Thymosin alpha1 & Pegylated Interferon-alpha2a

INTERVENTIONS:
Drug: Pegylated Interferon-alpha2a — 180 microgram s.c. injection weekly
  Arms: 1
Drug: Thymosin alpha1 & Pegylated Interferon-alpha2a — Pegylated interferon 180 microgram s.c. injection weekly Thymosin 1.6 mg s.c. injection twice per week
  Arms: 2

SUMMARY:
The purpose of this study is to determine the optimal treatment duration of antiviral therapy for chronic hepatitis B.

DETAILED DESCRIPTION:
Thymosin alpha1/interferon combination therapy has been known as an effective antiviral therapy for chronic hepatitis B. It is superior to interferon single therapy since the sustained viral response rate of combination therapy used to be about 70% compared with that of single interferon therapy(20%). Until now, the combination therapy including 6-month treatment of thymosin alpha1 has been as effective as 12-month treatment of thymosin alpha1. We hypothesized that thymosin alpha1 is an immune potentiator so, the shorter duration of thymosin alpha1 treatment might be as effective as the prolonged treatment duration.

In detail, we designed to perform this clinical study comparing the combination of pegylated interferon and thymosin alpha1 with pegylated interferon alone. Total treatment duration of both parallel groups will be 12 months, and the combination therapy will be lasted for the first 3 months followed by the next, ongoing pegylated interferon single therapy for 9 months.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive and anti-HBs negative for more than 6 months
* HBeAg positive
* HBV DNA titer more than 100,000 IU/mL
* serum ALT more than upper normal limit value, but no more than 10 times upper normal limit value

Exclusion Criteria:

* the history of antiviral therapy for chronic hepatitis B within the recent 6 months
* HAV IgM Ab + and/or HCV Ab + and/or HDV Ab and/or HIV Ab +
* the sign of decompensated liver disease
* the history of hemoglobinopathy, autoimmune hepatitis, alcoholic liver disease
* pregnant or lactating woman
* neutrophil count less than 1,500/mm3 or platelet count less than 90,000/mm3
* serum creatinine more than 1.5 times upper normal limit value
* the sign of alcoholic or drug addiction within the recent 1 year
* the history of psychotic disorder especially like depression
* immunologically mediated disease
* the history of esophageal varix
* the history of severe heart disease or respiratory disease
* the history of severe epilepsy or current use of antiepileptic drug
* the sign of malignancy or suggestive of malignancy or the history of malignancy, the recurrence rate within 2 years of which is more than 20%
* the history of systemic anticancer treatment including radiation therapy or immunotherapy including systemic corticosteroid
* the history of major organ transplantation
* the history of medically uncontrolled thyroid disease
* the history or sign of severe retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
HBeAg seroconversion, HBV DNA titer<20,000 IU/mL | 48 week and 96 week

SECONDARY OUTCOMES:
Normalization of serum ALT, loss of HBeAg and HBsAg, production of anti-HBs | 48 week and 96 week

CONTACTS AND LOCATIONS:
Overall Officials: Jung H Yoon, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Chongno-gu, South Korea